CLINICAL TRIAL: NCT04464356
Title: Application of Emergent Peripheral Mechanical Circulatory Support in Transcatheter Aortic Valve Replacement for 6 Patients
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-380
Record Dates: First submitted 2020-06-28; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Transcatheter Aortic Valve Replacement; Mechanical Circulatory Support
Keywords: transcatheter aortic valve replacement; mechanical circulatory support; cardiopulmonary bypass; ,extracorporeal membranous oxygenator

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: mechanical circulatory support — mechanical circulatory support: cardiopulmonary bypass, extracorporeal membrane oxygenation(ECMO), left ventricular assist device

SUMMARY:
Objective: To explore the experience of transcranial aortic valve replacement (TAVR) under emergency mechanical assisted circulation (MCS).Methods: A total of 6 patients who completed TAVR with the assistance of emergency MCS in the Second Affiliated Hospital of Zhejiang University School of Medicine from March 2013 to June 2019 were retrospectively analyzed.The management of perioperative mechanical assisted circulation, preoperative evaluation, intraoperative operation and postoperative situation of patients were summarized.

ELIGIBILITY:
Inclusion Criteria:

* TAVR patient, assisted by emergency peripheral MCS due to circulatory collapse during TAVR

Exclusion Criteria:

* patients presented mechanical complications such as massive hemorrhage, coronary artery occlusion or left ventricular rupture.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients assisted by emergency peripheral MCS during TAVR due to circulatory collapse.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
30-Day mortality rate | 30 days after TAVR procedure
  30-Day mortality rate

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No